CLINICAL TRIAL: NCT04313374
Title: Effective and Safe Morphine Dose for Patient Controlled Anesthesia in Supratentorial Craniotomies
Brief Title: Integrated Pulmonary Index and Opioid Based Patient Controlled Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Eren Fatma Akcil, SPECİALİST ANESTHESİOLOGİST, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cerrahpasa Neuroanaesthesia
Record Dates: First submitted 2018-02-28; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Brain Tumors
Keywords: Integrated pulmonary index, opioid side effects
MeSH Terms: conditions — Brain Neoplasms | interventions — Morphine; dexketoprofen trometamol; Acetaminophen

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Investigator
Masking Description: the patient, the investigator of the study will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Morphine PCA 1 mg (Active Comparator): The patient controlled analgesia device give 1mg morphine for each demand of the patient.
  Interventions: Drug: Morphine PCA 1 mg
- Morphine PCA 0,5 mg (Active Comparator): The patient controlled analgesia device give 0,5 mg morphine for each demand of the patient.
  Interventions: Drug: Morphine PCA 0,5 mg
- Placebo (Placebo Comparator): The patient controlled analgesia device give 2 mL serum physiologic for each demand of the patient.The Group 3 will take 50 mg dexketoprofen in the recovery room. Intra venous injections of dexketoprofen will repeat every 8 hours. If the VAS skore more than 4 the Group 3 patients will take 1 g paracetamol every 6 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Morphine PCA 1 mg — PCA will set to administer a bolus dose of 1 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours.
  Other Names: Morphine sulphate 1 mg
  Arms: Morphine PCA 1 mg
Drug: Morphine PCA 0,5 mg — PCA set to administer a bolus dose of 0.5 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours.
  Other Names: Morphine sulphate 0,5 mg
  Arms: Morphine PCA 0,5 mg
Drug: Placebo — the PCA will contain placebo
  Other Names: serum physiologic, dexketoprofen trometamol, paracetamol
  Arms: Placebo

SUMMARY:
An optimal analgesic therapy is very important for postoperative recovery. In recent years, several studies showed that the prevalence of the moderate to severe pain after craniotomy ranged from 69 to 87% of patients. The investigators showed that the use of morphine based patient controlled analgesia prevented moderate to severe postoperative pain in patients undergoing supratentorial craniotomy. Morphine related side effects such as sedation, miosis, respiratory depression, nausea and vomiting produce a general reluctance for their use in neurosurgery. Therefore, all patients were closely observed to detect opioid related side effects in the intensive care unit for 24 hours following surgery in our previous study. The Integrated Pulmonary Index (IPI) is a new tool that calculates respiratory and hemodynamic parameters noninvasively. In the present study the investigators will use different doses of morphine based patient-controlled analgesia and the IPI system to determine more effective and safer morphine dose for postoperative analgesia following supratentorial craniotomy.

DETAILED DESCRIPTION:
An optimal analgesic therapy is very important for postoperative recovery. In recent years, several studies showed that the prevalence of the moderate to severe pain after craniotomy ranged from 69 to 87% of patients. In our previous study, the investigators showed that the use of morphine based patient controlled analgesia prevented moderate to severe postoperative pain in patients undergoing supratentorial craniotomy. Morphine related side effects such as sedation, miosis, respiratory depression, nausea and vomiting produce a general reluctance for their use in neurosurgery. Therefore, all patients were closely observed to detect opioid related side effects in the intensive care unit for 24 hours following surgery in our previous study. The Integrated Pulmonary Index (IPI) is a new tool that calculates respiratory and hemodynamic parameters noninvasively. In the present study The investigators will use different doses of morphine based patient-controlled analgesia and the IPI system to determine more effective and safer morphine dose for postoperative analgesia following supratentorial craniotomy.

90 patients will randomize in 3 groups following supratentorial craniotomy. All patients will previously instruct on the patient-controlled analgesia pumps (Abbott Provider, Chicago, USA) and visual analogue scale (VAS) from 0 to 10, with 0 being no pain and 10 being the worst pain imaginable. All patients will use patient-controlled analgesia pumps for 24 hours following supratentorial craniotomy. In the Group 1 the patient-controlled analgesia pump will set to administer a bolus dose of 1 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours. In the Group 2 the patient-controlled analgesia pump will set to administer a bolus dose of 0.5 mg morphine on demand with a lockout period of 10 minutes and maximum 20 mg for 4 hours. In the Group 3 the patient-controlled analgesia pump will contain placebo. The Group 3 will take 50 mg dexketoprofen in the recovery room. Intra venous injections of dexketoprofen will repeat every 8 hours. If the VAS score will more than 4 the Group 3 patients will take 1 g paracetamol every 6 hours.

All patients will be observed by the Integrated Pulmonary Index (IPI). It is a new device that provides to recognise in a patients respiratory status. This software tool is a single index value ranging from 1 to 10 based on 4 physiological parameters: end tidal carbon dioxide, respiratory rate, oxygen saturation, pulse rate. Patients will asses at 10th minute, 1, 2, 6, 12, and 24 hours postoperatively. Sedation will evaluate according to Ramsay score 20. VAS scores, total morphine consumption, Ramsay score, blood pressure, heart rate and respiratory rate, the IPI score will record at each time pain will evaluate. Postoperative side effects, including rash, pruritus, nausea and vomiting will record at the same intervals and defined by a scale with 0 = absent or 1 = present. Moreover the lowest IPI score, the apnea count (longer than 30 seconds) and the count of the desaturation events will record in the postoperative 24 hours.

The 3 Groups will compare with respect to VAS scores, morphine consumption, IPI scores, the apnea count, the desaturation events and morphine related side effects during the 24 hours following supratentorial craniotomy.

ELIGIBILITY:
Inclusion Criteria: , brain tumors, elective supratentorial craniotomies,

* Conscious patients
* Elective supratentorial craniotomies
* ASA I-III

Exclusion Criteria:

* Unconscious postoperatively
* Chronic pain
* Opioid, dexketoprofen or paracetamol allergy
* Delirium
* Renal insufficiency
* Alcohol, opioid dependency
* Transsphenoidal pituitary surgery

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Integrated pulmonary index system | 24 hour postoperatively
  Integrated pulmonary index system will be used to determine more effective and safer morphine dose for postoperative analgesia following supratentorial craniotomy. This software tool is a single index value ranging from 1 to 10 based on 4 physiological parameters: end tidal carbon dioxide, respiratory rate, oxygen saturation, pulse rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Tunali, Professor, Study Director — Cerrahpasa Medical School
Locations (1):
- Istanbul University Cerrahpasa Medical School, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Thibault M, Girard F, Moumdjian R, Chouinard P, Boudreault D, Ruel M. Craniotomy site influences postoperative pain following neurosurgical procedures: a retrospective study. Can J Anaesth. 2007 Jul;54(7):544-8. doi: 10.1007/BF03022318. PMID 17602040
- [Background] Mordhorst C, Latz B, Kerz T, Wisser G, Schmidt A, Schneider A, Jahn-Eimermacher A, Werner C, Engelhard K. Prospective assessment of postoperative pain after craniotomy. J Neurosurg Anesthesiol. 2010 Jul;22(3):202-6. doi: 10.1097/ANA.0b013e3181df0600. PMID 20479664